CLINICAL TRIAL: NCT01314495
Title: A Randomized, Double Blind, Placebo Controlled Clinical Trial to Evaluate the Efficacy of Abatacept Costimulatory Blockade in the Treatment of Alopecia Totalis/Universalis
Brief Title: Abatacept Costimulatory Blockade in the Treatment of Alopecia Totalis/Universalis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Halt in funding
Sponsor: Julian M. Mackay-Wiggan (Other)
Responsible Party: Sponsor-Investigator, Julian M. Mackay-Wiggan, Assistant Clinical Professor of Dermatology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAI1530
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Alopecia Totalis/Universalis
Keywords: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abatacept (Active Comparator): Abatacept administered as a 30 minute intravenous infusion
  Interventions: Drug: Abatacept
- Inactive infusion (Placebo Comparator): Placebo will be administered as a 30 minute intravenous infusion.
  Interventions: Drug: Inactive infusion

INTERVENTIONS:
Drug: Abatacept — Abatacept will be administrated as a 30 minute intravenous infusion.
  Arms: Abatacept
Drug: Inactive infusion — Placebo will be administered as a 30 minute intravenous infusion.
  Arms: Inactive infusion

SUMMARY:
Will Abatacept reduce priming of the hair follicle specific T cells and thereby reduce hair follicle associated infiltration and improve hair growth.

This is a double blind placebo controlled study to test the safety and efficacy of Abatacept in the treatment of 64 subjects diagnosed with alopecia totalis or alopecia universalis. Subjects will be randomized 1:1 to the placebo or treatment arm and will receive 6 months of treatment with the study medication or placebo, followed by a 6 month observational period.

DETAILED DESCRIPTION:
Alopecia Areata is a common autoimmune disease, affecting 1% of the general population resulting from autoimmune attack on the hair follicles and usually presents with patchy hair loss. One third of these patients will experience spontaneous remissions within the first year. However many patients will develop waxing and waning disease with some progressing to alopecia totalis (total scalp hair loss) or alopecia universalis (loss of all body hair). This population that suffers from a disfiguring disease represents a significant unmet medical need. Alopecia totalis/universalis seldom, if ever, remits spontaneously or with current treatment and is classified by the FDA as an Orphan Indication.

There is no FDA approved drug for alopecia areata. A recent Cochrane report concluded that there was no evidence based support for any intervention in this disease. Standard of care remains observation for mild disease and lesional/oral steroids for more advanced cases.

Abatacept is a soluble human fusion protein that selectively modulates the costimulatory signal required for full T-cell activation. It is approved for the treatment of moderately to severely active rheumatoid arthritis. It is also approved for the treatment of moderately to severely active polyarticular juvenile idiopathic arthritis in children 6 years of age or older. Abatacept is a lyophilized powder administered as a 30 minute intravenous infusion. Dosage, as in rheumatoid arthritis, is weight based and is fixed throughout the course of treatment. Abatacept or placebo will be administered as a 30 minute intravenous infusion at baseline, weeks 2, 4, and every 4 weeks for 5 cycles (weeks 8, 12, 16, 20) for a total treatment period of 6 months. There will be a 6 month observational period following the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 75 years of age.
* Must have a diagnosis of alopecia totalis or alopecia universalis
* Must have >75% total scalp hair loss at baseline as measured using the SALT score.
* Duration of hair loss must be between 3 to 12 months.
* There may be no evidence of regrowth present at baseline.
* Subjects may be naïve to treatment or unresponsive to intralesional (IL) steroids or other treatments for alopecia areata.
* Must be willing to avoid live vaccines while on the study medication, and within 3 months of its discontinuation.

Exclusion Criteria:

* Patients with a history of or active skin disease on the scalp such as psoriasis or seborrheic dermatitis.
* Patients in whom the diagnosis of alopecia areata is in question.
* Patients with active medical conditions or malignancies (except adequately treated basal or squamous cell carcinoma) that in the opinion of the investigator would increase the risks associated with study participation, including patients with a history of recurrent infections.
* Patients who monitor their blood glucose levels using glucose dehydrogenase pyrrologuinolinequinone (GDH-PQQ) test strips. Blood glucose monitoring using other methods that do not react with maltose, such as the glucose dehydrogenase nicotine adenine dinucleotide (GDH-NAD), glucose oxidase, or glucose hexokinase test methods are permitted.
* Patients taking TNF antagonists or other biological therapy such as anakinra.
* Women of childbearing potential who are unable or unwilling to use two forms of birth control for the study duration.
* Women who are pregnant or nursing.
* Patients known to be HIV or hepatitis B or C positive.
* Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening.
* Patients with latent Mycobacterium tuberculosis infection as indicated by a positive Purified Protein Derivative [PPD] skin test. Subjects with a positive PPD skin test and documented completion of treatment per standard medical practice for latent TB are eligible. Subjects with a positive PPD skin test and not treated or no documentation of completion of treatment are ineligible.
* History of incompletely treated Mycobacterium tuberculosis infection as indicated by:
* Subject's medical records documenting incomplete treatment for Mycobacterium tuberculosis
* Subject's self-reported history of incomplete treatment for Mycobacterium tuberculosis
* Patients with evidence of infection or skin cancer in the treated areas.
* Patients with history or evidence of hematopoietic abnormality.
* Patients with history of immunosuppression or history of recurrent serious infections.
* Patients with a history or likely diagnosis of COPD
* Patients unwilling or unable to discontinue treatments known to affect hair regrowth in alopecia areata.
* Patients who have been treated with intralesional steroids, systemic steroids, anthralin, squaric acid, DPCP (diphenylcycloprophenone), protopic, minoxidil or other medication which in the opinion of the investigator may affect hair regrowth within one month of the baseline visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The study's primary endpoint will be the proportion of responders after 6 months of treatment, defined as 50% or greater hair re-growth from baseline as assessed by Severity of Alopecia Tool (SALT) score at week 24. | 24 weeks
  The study's primary endpoint of this intent to treat trial will be the proportion of responders in the treated compared to the control group after 6 months of treatment, defined as 50% or greater hair re-growth from baseline as assessed by Severity of Alopecia Tool (SALT) score at week 24. This is a relatively strict definition for defining responders and non-responders and was chosen to minimize responses in the 'vehicle' arm, in which fewer than 10% are expected to achieve this magnitude of hair re-growth spontaneously.

SECONDARY OUTCOMES:
Percent hair regrowth from baseline determined by SALT at weeks 4, 8, 12, 20, and 24 during treatment phase and at weeks 30, 36, 42 and 48 during the observational phase. | 24 weeks of treatment and 18 weeks observational phase
  As secondary endpoints, efficacy will be measured by changes in hair re-growth as a continuous variable as determined by physical exam and photography, as well as subject and physician global evaluation scores. To assess the durability of responses, subjects will continue to be followed for an additional 6 months post treatment. All subjects will be assessed for safety at each study visit for incidence and severity of adverse effects (AE) and incidence of treatment emergent laboratory abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Mackay-Wiggan, MD, MS, Principal Investigator — Columbia University; Angela Christiano, PhD, Study Director — Columbia University